CLINICAL TRIAL: NCT02910479
Title: Phase 1 Study Evaluating the Relevance and Reliability of Gastrointestinal Temperature Measurements From a New Device (E-celsius)
Brief Title: Study Evaluating the Relevance and Reliability of Gastrointestinal Temperature Measurements From a New Device (E-celsius)
Acronym: e-TEMP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); La Région Basse-Normandie (Other); Université de Caen Normandie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-167
Record Dates: First submitted 2016-03-17; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers
Keywords: Body Temperature; Thermometers
MeSH Terms: interventions — Thermometers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temperature measurements with 4 devices (Experimental): temperature measurements with e-device Celsius, esophageal probe and a rectal probe and vital sense capsule
  Interventions: Device: E-Celsius thermometer; Device: Rectal thermometer; Device: Esophageal thermometer; Device: Vital sense capsule thermometer

INTERVENTIONS:
Device: E-Celsius thermometer — comparison of temperature between e-celsius and thermometer, rectal thermometer, esophageal thermometer, vital sense capsule thermometer
Device: Rectal thermometer
Device: Esophageal thermometer
Device: Vital sense capsule thermometer

SUMMARY:
E-Celsius device used for measuring the gastrointestinal temperature is composed of an ingestible capsule measuring the temperature as well as a transportable module receiving data from the capsule. This device allows to measure the body temperature (± 0.2 ° C) during transit of the pill in the digestive tract to a maximum sampling frequency of 30 seconds. The main risks related to such devices are related to biocompatibility (in materials used for the capsule shell, or level of contamination of the gastrointestinal environment due to a defect in the plastic envelope the pill or a lack of hygiene, previously tested in clinical trials; see section 10.2).

It will compare conventional methods of estimating the central temperature continuously with gastrointestinal data obtained from the e-Celsius device. The main objective of the research is to validate the extent of gastrointestinal temperature obtained from the device under test consists of an ingestible electronic capsule and a data reception monitor.

Secondary objectives will be pursued:

* Assess the effects of ingestion of cold drinks on temperature readings taken via e-device Celsius, esophageal probe and a rectal probe.
* Explore the thermal homogeneity of the digestive tract.
* Evaluate the internal memory of the capsule and its data forwarding capacity. This protocol will also measure the reliability of the measurement system while comparing it to the standards used by health staff today.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers male or female (18 to 59 years inclusive)
* Signed the informed consent.
* Affiliated to the social security scheme
* French speaker

Exclusion Criteria:

* Subject having started or stopped during the 15 days preceding the inclusion visit one of the following treatments: antidepressants, anxiolytics, antiparkinsonian agents, neuroleptics.
* Subject having taken over the previous 7 days a drug to treat irritable bowel syndrome (antispasmodic, etc ...) or constipation (laxative)
* Subject with known food allergies
* Subject undergoing surgery for colon surgery
* Subject with an organic occlusion
* Subject with known abnormal liver or renal function
* Subject participating in another clinical study within a month before the inclusion visit.
* A person with a bodyweight under 40 kg
* Any person with obstruction (known or suspected) of the gastrointestinal tract, including people with diverticula (folds) intestinal or intestinal inflammation known.
* People with a BMI greater than or equal to 30.
* People under guardianship
* People who have or had known swallowing disorders
* People who have to undergo an MRI or to be subjected to a strong magnetic field programmed during the transit of the capsule
* Persons equipped with a pacemaker
* People with diabetes or with diabetic history
* People with heave
* The detainees
* Pregnant women
* People with nasal septum deviation
* People with against-indications to the placement of an esophageal tube: people who carry chronic esophageal pathology (eg, gastroesophageal reflux treated, hiatal hernia,)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
body temperature | from baseline to 36 hours every minute
  comparisons between device e-Celsius, esophageal probe and a rectal probe

SECONDARY OUTCOMES:
body temperature during ingestion of cold drinks | baseline
  Assess the effects of ingestion of cold drinks on temperature readings taken via e-device Celsius, esophageal probe and a rectal probe
temperature of the digestive tract | from baseline to 36 hours every minute
  Explore the thermal homogeneity of the digestive tract
number of lost data | from baseline to 36 hours every minute
  The capacity of the for each measurements method to store temperature data in the internal memory and send it to the receiver when the it is in the receiving area.
reliability of measurements | from baseline to 36 hours every minute
  reliability of the measurement system while comparing it to the standards used by health staff today

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France